CLINICAL TRIAL: NCT03578484
Title: Breast Aesthetics by Three Dimensional Measures - A Transatlantic Evaluation of Beauty Ideals Using 3D Scanning and Mammometrics.
Brief Title: Breast Aesthetics by Three Dimensional Measures
Status: Active, not recruiting | Type: Observational
Sponsor: Sykehuset Telemark (Other Government)
Collaborators: M.D. Anderson Cancer Center (Other); University College of Southeast Norway (Other); Skintech A/S (Unknown); Canfield Inc (Unknown); Oslo University Hospital (Other); Karolinska Institutet (Other); University of Helsinki (Other)
Responsible Party: Sponsor
Other Study IDs: 44059 / 3 / MSS
Record Dates: First submitted 2018-04-25; First posted 2018-07-06 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer
Keywords: Breast Aesthetics; 3D scanning; Aesthetic rating; Cultural Differences Aesthetics; Mammometrics
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Volunteer female subjects: Females age 18-35 years of age. 3D breast scan will be performed and followed over 15 years. No therapeutic interventions will be performed.
  Interventions: Diagnostic Test: Aesthetic assessment 3D breast scanning

INTERVENTIONS:
Diagnostic Test: Aesthetic assessment 3D breast scanning — Vectra TM - Canfield Inc breast scan. 3D digital photography scan.

SUMMARY:
Traditionally the measures of the optimally aesthetic breast have been assumed to be static and to represent universal values (1). Measures developed for optimal aesthetic results in breast reduction were derived from brassiere patterns and then applied universally (2). These early and important papers still strongly influence the view of the aesthetics of the breast despite the lack of individualisation and proportion.

To create satisfying results for specific patients, optimal proportions angles and relative measures are needed for each patient. The study will clarify theses measures and provide important guidelines for surgeons.The data will also help define optimal proportional aesthetics in the individual patient.

The concept of universal beauty is unrealistic. It has always been taken for granted that aesthetic values from all cultures are similar. Using 3D scanning on volunteers of youthful age offers a complex set of data that may distinguish fine differences in aesthetic ideals in different cultures.

Little is known about how life events and life-style factors affect breast aesthetics.

To follow a population with 3D scans over 5, 10 and 15 years will allow aesthetic ratings to be correlated with life events such as pregnancy, childbirth, breast-feeding and life style factors such as smoking.

The study will improve the understanding of breast aesthetics in general, in different cultures and in relation to life events and life style factors. No similar studies have previously been performed.

DETAILED DESCRIPTION:
Aims for the study:

To identify aesthetic factors that contribute to overall beauty and aesthetics of the breast.

To identify proportions and measures of the most aesthetically pleasing breast and also of the least appealing breast. This will provide a guideline and a map for the reconstructive breast surgeon in what to aim for and what to avoid in the breast reconstructive process.

To identify cultural differences in the perception of beauty.

Aims for the longitudinal part of the study:

To identify lifestyle and life event factors that independently influences the progression of cosmetic ratings and 3D measurements of the breast over 5, 10 and 15 years.

To identify trends and differences in aesthetic ratings of the same 3D scans over time.

Data collection:

At the initial and all following controls of the study a short patient interview will be conducted to obtain the following information:

Subject demographics:

Age, Race, Previous Medical History, Number of Childbirths, Breast feeding - how many children - how many months per child, Surgeries of the breast, Surgeries of the chest wall, Weight, Height, Bra Size, Sports bra use - always - during sports - rarely - never, Smoking, alcohol, Occupation, Physical activity

Measures of the breast will be obtained by 3D scanning.

Rating of the 3D scans will be performed by eight assigned teams:

10 Plastic Surgeons from Scandinavia, 10 Plastic Surgeons from Texas, 10 Scandinavian nurses without formal aesthetic or plastic surgery training, 10 Nurses and/or Physician assistants from the USA without formal aesthetic or plastic surgery training, 10 Medical Students from Texas, 10 Medical Students from Scandinavia, 10 Nursing Students from Texas, 10 Nursing Students from Scandinavia

The 3D scans will be aesthetically rated by independent evaluators on a scale from 1-5. The vertical split plane and the horizontal split plane as defined by Tepper et al (8) in mammometrics will be used to subdivide the breast into aesthetic units.

A separate rating will be obtained for each breast:

Lower pole 1-5, Upper pole 1-5, Medial pole 1-5, Lateral pole 1-5, Nipple position 1-5, Areola color 1-5, Areola size 1-5, Breast footprint position, Overall score

Also both breasts together will be scored regarding:

Intermammary distance / breast cleft, symmetry, overall bilateral score

Data Storage:

The data will be stored for 16 years. The data will be stored in a password -protected computer with firewall protection. The data will be stored in a locked safe.

Statistics:

We will use descriptive statistics such as mean and standard deviation. Various subgroup analyses may occur - continuous variables will be compared using the two sample T-test and parametric variables will be compared using chi-squared analysis or Fischer's exact test. Univariate and multivariate regression models will be used to analyze for confounding factors.

The statistical calculations will be performed in Norway at the Dept of statistics at Rikshospitalet Oslo and/or in collaboration with MD Anderson Cancer Center in Texas, USA.

The rating-system for aesthetics will be tested for reliability. Ten raters will be rating 30 of the same 3D scans twice with a 2 week interval.

Calculation of necessary number of participating women (n) as determined in collaboration with the Dept of Statistics Oslo University:

In the present study a mean score of "overall score bilateral breasts" will be compared in 10 American (Group 1, 3, 5, 7) and 10 Scandinavian/Norwegian (Group 2, 4, 6, 8) plastic surgeons/nurses/medical students/nursing students. We define a mean "overall score bilateral breasts" score difference of at least 0.5 to be a difference of statistical significance. Significance will be defined as p = 0.05. In order to perform a power calculation we need an estimate of the standard deviation (SD) of the scoring of "overall score bilateral breasts" within each group. However such estimates are not available in the literature. We therefore will use the following procedure to calculate (n):

Step 1: Include 10 women and measure average score on "overall score bilateral breasts" for each plastic surgeon. Then calculate SD for each of the average scores in each group. Then we will use these estimates of SD in a power calculation, and calculate the (n) associated with a test power of 80% as per Sandvik.

Our preliminary estimation of power is 150 patients. The somewhat high number is due to potential drop out rates for the longitudinal arm of the study.

Organisation:

Principal Investigator and Conceptual Author: LJ Sandberg Telemark Hospital Trust, Dept of Plastic Surgery, Norway

Collaborators:

Senior author: JC Selber MD Anderson Cancer Center, USA Other authors in random order: G Reece MD Anderson Cancer Center, USA; K Kloster Jensen Telemark Hospital Trust Dept of Plastic Surgery; T Bernklev Telemark Hospital Trust, Dept of Research, Norway; L Sandvik Oslo University, Dept of Statistics, Norway; G Gunnarson Telemark Hospital Trust, Dept of Plastic Surgery, Norway; E Berg Telemark Hospital Trust, Dept of Plastic Surgery, Norway; K Tønseth, Oslo University Hospital, Dept of Plastic Surgery, Norway; HP Gullestad, Oslo University Hospital, Dept of Plastic Surgery, Norway; M Halle Dept of Plastic Surgery, Karolinska Institute Sweden; Å Edsander Nord Dept of Plastic Surgery, Karolinska Institute Sweden; A Höckerstedt Dept of Plastic Surgery, University of Helsinki, Finland; S Kauhanen Dept of Plastic Surgery, University of Helsinki, Finland; E Holm Hansen University Southeast Norway, Norway; Karin Berntsen University Southeast Norway, Norway; Plastic Surgical Department of Statistics at MD Anderson Cancer Center , USA; Department of Statistics at Oslo University, Norway

Canfield Inc / Skintech are not active partners in the project, just partners supplying technology and support. The name of the 3D Vectra system will be used in the paper to scientifically describe the study. Canfield Inc will be mentioned in the Method section of the study as contributing to the study and any conflicts of interests will be disclosed in all and any presentations and publications. No funds have been received from Canfield Inc. Canfield Inc has allowed use of the Vectra 3D camera in the study without any demands or charges.

Clinical Importance:

Aesthetic measures are the basis of all plastic surgical breast procedures and this study will have a major influence on all of plastic surgical procedures of the breast - particularly breast reconstruction. Determining a difference between aesthetic ratings in different cultures would further stress the concept of "beauty lying in the eye of the beholder" and that beauty concepts have to be adapted to the individual and not the other way around. Beauty is not one strict measure, but a range of measures and proportions adapted to the individual subject. The use of 3D scanning is a new technique that offers superior quality documentation and preoperative analysis. The study will further define 3D scanning as a new standard for aesthetic breast evaluations.

In the long term follow up the factors affecting aesthetic ratings over time (aging of the breast), such as smoking, would be revealed. This could further allow life style choices to be made by patients promoting breast aesthetics and hopefully health in general.

ELIGIBILITY:
Inclusion Criteria:

* The study will be based on female volunteers between the ages of 18 and 35 of all ethnic backgrounds.

Exclusion Criteria:

* Patients with breast cancer treatment, removal of non-malignant masses, trauma, burns or dermatological diagnoses involving the breast are excluded from the study.

Ages: 18 Years to 35 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Only the female breast aesthetics are evaluated.
Study Population: The study will be based on female volunteers between the ages of 18 and 35 of all races. This age range incorporates early to late youth. It also allows for sequential follow up. Patients with breast cancer treatment, removal of non-malignant masses, trauma, burns or dermatological diagnoses involving the breast were excluded from the study. Subjects with cosmetic surgery will be allowed to participate in the study. Volunteers will be recruited from nursing staff at Telemark Health Trust, nursing students from University Southeast Norway in Porsgrunn Norway.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2016-05-13 (Actual); Primary Completion 2032-03-20 (Estimated); Study Completion 2032-03-20 (Estimated)

PRIMARY OUTCOMES:
Breast aesthetic score in Scandinavia | 5 years
  Using a rating system developed by Sandberg and Selber for this project, each individual breast (left and right) will be scored according to aesthetic aspects. A score ranging from 1 lowest to 5 highest will be given by the rater. The parameters rated will be breast size, breast width, breast height, breast position, nipple position, nipple shape, nipple color and breast shape.
  The score will be the outcome measure for the most pleasant aesthetics.
Breast measures in centimeters and degrees in Scandinavia | 5 years
  The highest and lowest scored breasts will be measured. Anatomic measures of the breast between fiduciary points, such as distance the nipple and the sternal notch in centimeters. Also measures of angles between the midline and nipple position measured in degrees. Also measures of curvatures in degrees and vectors. The measures will be performed digitally on the 3D scans obtained by the Vectra system for 3D scanning using the software developed by Canfield Inc.
  This will be the outcome measure in centimeters, degrees and proportions.
Breast aesthetic score in USA | 5 years
  Using a rating system developed by Sandberg and Selber for this project, each individual breast (left and right) will be scored according to aesthetic aspects. A score ranging from 1 lowest to 5 highest will be given by the rater. The parameters rated will be breast size, breast width, breast height, breast position, nipple position, nipple shape, nipple color and breast shape.
  The score will be the outcome measure for the most pleasant aesthetics in the USA.
Breast measures in centimeters and degrees in USA | 5 years
  The highest and lowest scored breasts will be measured. Anatomic measures of the breast between fiduciary points, such as distance the nipple and the sternal notch in centimeters. Also measures of angles between the midline and nipple position measured in degrees. Also measures of curvatures in degrees and vectors. The measures will be performed digitally on the 3D scans obtained by the Vectra system for 3D scanning using the software developed by Canfield Inc.
  This will be the outcome measure in centimeters, degrees and proportions for USA.

SECONDARY OUTCOMES:
Breast measures in centimeters and degrees changes at 5 years | 10 years
  The highest scored breasts will be measured. Anatomic measures of the breast between fiduciary points, such as distance the nipple and the sternal notch in centimeters. Also measures of angles between the midline and nipple position measured in degrees. Also measures of curvatures in degrees and vectors. The measures will be performed digitally on the 3D scans obtained by the Vectra system for 3D scanning using the software developed by Canfield Inc.
  This will be the outcome measure in centimeters, degrees and proportions to detect change after 5 years.
Breast measures in centimeters and degrees changes at 10 years | 15 years
  The highest scored breasts will be measured. Anatomic measures of the breast between fiduciary points, such as distance the nipple and the sternal notch in centimeters. Also measures of angles between the midline and nipple position measured in degrees. Also measures of curvatures in degrees and vectors. The measures will be performed digitally on the 3D scans obtained by the Vectra system for 3D scanning using the software developed by Canfield Inc.
  This will be the outcome measure in centimeters, degrees and proportions to detect change after 10 years.
Breast measures in centimeters and degrees changes at 15 years | 16 years
  The highest scored breasts will be measured. Anatomic measures of the breast between fiduciary points, such as distance the nipple and the sternal notch in centimeters. Also measures of angles between the midline and nipple position measured in degrees. Also measures of curvatures in degrees and vectors. The measures will be performed digitally on the 3D scans obtained by the Vectra system for 3D scanning using the software developed by Canfield Inc.
  This will be the outcome measure in centimeters, degrees and proportions to detect change after 15 years.
Change in breast aesthetic score at 5 years | 10 years
  Using a rating system developed by Sandberg and Selber for this project, each individual breast (left and right) will be scored according to aesthetic aspects. A score ranging from 1 lowest to 5 highest will be given by the rater. The parameters rated will be breast size, breast width, breast height, breast position, nipple position, nipple shape, nipple color and breast shape.
  The score will be the outcome measure for the change of aesthetics over 5 years.
Change in breast aesthetic score at 10 years | 15 years
  Using a rating system developed by Sandberg and Selber for this project, each individual breast (left and right) will be scored according to aesthetic aspects. A score ranging from 1 lowest to 5 highest will be given by the rater. The parameters rated will be breast size, breast width, breast height, breast position, nipple position, nipple shape, nipple color and breast shape.
  The score will be the outcome measure for the change of aesthetics over 10 years.
Change in breast aesthetic score at 15 years | 16 years
  Using a rating system developed by Sandberg and Selber for this project, each individual breast (left and right) will be scored according to aesthetic aspects. A score ranging from 1 lowest to 5 highest will be given by the rater. The parameters rated will be breast size, breast width, breast height, breast position, nipple position, nipple shape, nipple color and breast shape.
  The score will be the outcome measure for the change of aesthetics over 15 years.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Johan M Sandberg, MD, FACS, Principal Investigator — STHF
Locations (2):
- Norway (2):
  - Sykehuset Telemark, Skien, Telemark
  - Oslo University Hospital, Oslo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] PENN J. Breast reduction. Br J Plast Surg. 1955 Jan;7(4):357-71. doi: 10.1016/s0007-1226(54)80046-4. No abstract available. PMID 13230442
- [Result] WISE RJ. A preliminary report on a method of planning the mammaplasty. Plast Reconstr Surg (1946). 1956 May;17(5):367-75. doi: 10.1097/00006534-195605000-00004. No abstract available. PMID 13335513
- [Result] Loughry CW, Sheffer DB, Price TE Jr, Lackney MJ, Bartfai RG, Morek WM. Breast volume measurement of 248 women using biostereometric analysis. Plast Reconstr Surg. 1987 Oct;80(4):553-8. doi: 10.1097/00006534-198710000-00013. PMID 3659165
- [Result] Loughry CW, Sheffer DB, Price TE, Einsporn RL, Bartfai RG, Morek WM, Meli NM. Breast volume measurement of 598 women using biostereometric analysis. Ann Plast Surg. 1989 May;22(5):380-5. doi: 10.1097/00000637-198905000-00002. PMID 2729845
- [Result] Smith DJ Jr, Palin WE Jr, Katch VL, Bennett JE. Breast volume and anthropomorphic measurements: normal values. Plast Reconstr Surg. 1986 Sep;78(3):331-5. doi: 10.1097/00006534-198609000-00008. PMID 3737757
- [Result] Losken A, Seify H, Denson DD, Paredes AA Jr, Carlson GW. Validating three-dimensional imaging of the breast. Ann Plast Surg. 2005 May;54(5):471-6; discussion 477-8. doi: 10.1097/01.sap.0000155278.87790.a1. PMID 15838205
- [Result] Tepper OM, Small K, Rudolph L, Choi M, Karp N. Virtual 3-dimensional modeling as a valuable adjunct to aesthetic and reconstructive breast surgery. Am J Surg. 2006 Oct;192(4):548-51. doi: 10.1016/j.amjsurg.2006.06.026. PMID 16978973
- [Result] Tepper OM, Unger JG, Small KH, Feldman D, Kumar N, Choi M, Karp NS. Mammometrics: the standardization of aesthetic and reconstructive breast surgery. Plast Reconstr Surg. 2010 Jan;125(1):393-400. doi: 10.1097/PRS.0b013e3181c4966e. No abstract available. PMID 20048631
- [Result] Rohrich RJ, Bolden K. Ethnic rhinoplasty. Clin Plast Surg. 2010 Apr;37(2):353-70. doi: 10.1016/j.cps.2009.11.006. PMID 20206751
- [Result] Li Z, Unger JG, Roostaeian J, Constantine F, Rohrich RJ. Individualized Asian rhinoplasty: a systematic approach to facial balance. Plast Reconstr Surg. 2014 Jul;134(1):24e-32e. doi: 10.1097/PRS.0000000000000294. PMID 25028852